CLINICAL TRIAL: NCT06028594
Title: An Expanded Access Program of Pozelimab and Cemdisiran Combination Therapy in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Compassionate Use of Pozelimab and Cemdisiran Combination Therapy in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: No longer available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R3918-PNH-2238
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Pozelimab — Subcutaneous (SC) administration
  Other Names: REGN3918
Drug: Cemdisiran — Subcutaneous (SC) administration
  Other Names: ALN-CC5

SUMMARY:
This program is designed to provide access to pozelimab and cemdisiran and document the long-term safety of pozelimab and cemdisiran combination therapy in patients with paroxysmal nocturnal hemoglobinuria (PNH). PNH is a rare immune disease that causes red blood cells in your body to break apart.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients who have completed either the end of treatment visit of the open-label treatment period or open-label extension period in one of the following parent studies:

   * An Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of Pozelimab and Cemdisiran Combination Therapy in Patients with Paroxysmal Nocturnal Hemoglobinuria (R3918-PNH-2050 [NCT05744921])
   * A Randomized, Open-Label, Two-Arm Study to Evaluate the Safety, Efficacy, and Pharmacodynamic Effects of Pozelimab and Cemdisiran Combination Treatment in Patients with Paroxysmal Nocturnal Hemoglobinuria Who Have Received Pozelimab Monotherapy (R3918-PNH-2092 [NCT04811716])
   * A Single Arm, Open-Label Study to Assess the Safety, Efficacy, and Pharmacodynamic Effects of Pozelimab and Cemdisiran Combination Therapy in Patients with Paroxysmal Nocturnal Hemoglobinuria Who Switch from Eculizumab Therapy (R3918-PNH-20105 [NCT04888507]). Note: In some countries, patients that would normally enter into the R3918-PNH-2050 (NCT05744921) parent study before entering this expanded access program, may be given the opportunity to skip R3918-PNH-2050 (NCT05744921) and go straight into this expanded access program, with Regeneron's permission
2. Patients who have been enrolled in R3918-PNH-2022 (NCT05131204), with Regeneron's permission
3. Willing and able to comply with clinic visits and related standard-of-care procedures
4. With Regeneron's permission, patients who have been enrolled in other PNH studies as appropriate

Key Exclusion Criteria:

1. Significant history or concerns of non-compliance that could impact the patient's safety per the treating physician
2. Any new condition or worsening of an existing condition which, in the opinion of the treating physician, would make the patient unsuitable for enrollment or could interfere with the patient participating in or completing the program

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult